CLINICAL TRIAL: NCT00023504
Title: Evaluation of Immune Response to Vaccines in Primary Immune Disorders
Brief Title: Antibody Production in Immune Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow/Insufficient accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 010226; 01-I-0226
Record Dates: First submitted 2001-09-07; First posted 2001-09-10 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Primary Immune Deficiency
Keywords: Antibody; Vaccination
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pneumococcal Vaccine (Active Comparator): To determine the function of T and B cells in vivo using Pneumococcal vaccine immunization in patients with known or suspected immune disorders.
  Interventions: Biological: Pneumovax; Biological: Prevnar; Biological: Tetanus diphtheria toxoid
- Rabies Vaccine (Active Comparator): To determine the function of T and B cells in vivo using Rabies vaccine immunization in patients with known or suspected immune disorders.
  Interventions: Biological: Rabavert

INTERVENTIONS:
Biological: Pneumovax — To determine the function of T and B cells in vivo using immunizations in patients with known or suspected immune disorders.
  Arms: Pneumococcal Vaccine
Biological: Rabavert — To determine the function of T and B cells in vivo using immunizations in patients with known or suspected immune disorders.
  Arms: Rabies Vaccine
Biological: Prevnar — To determine the function of T and B cells in vivo using immunizations in patients with known or suspected immune disorders.
  Arms: Pneumococcal Vaccine
Biological: Tetanus diphtheria toxoid — To determine the function of T and B cells in vivo using immunizations in patients with known or suspected immune disorders.
  Arms: Pneumococcal Vaccine

SUMMARY:
This study will evaluate immune function in people with a known or suspected immune disorder. It will determine participants immune response to vaccines by measuring blood antibody levels after vaccination.

Patients enrolled in a NIH protocol involving immune reconstitution (bone marrow transplantation or gene therapy) for a known or suspected primary immune disorder may be eligible for this study.

Participants may be asked to have more than one vaccine, based on their age, use of IVIG, past immunization history and underlying immune problem. The possible vaccinations include:

Rabies vaccine

Diphtheria and tetanus booster

23 valent pneumococcal polysaccharide vaccine

Pneumococcal 7-valent conjugate vaccine

The diphtheria, tetanus, pneumococcus and rabies vaccines are approved by the Food and Drug Administration (FDA) and used routinely to protect against disease.

Study participants will have a blood sample drawn before vaccination. The number of additional samples collected will vary according to the vaccines administered; 1 for rabies; 1 for tetanus; and 1 to 2 for the pneumococcal vaccines. Each sample will be up to 5 teaspoonfuls. Participation in the study may last up to a year, depending on the blood sampling scheduling

DETAILED DESCRIPTION:
The purpose of this study is to evaluate immune responses to vaccines in subjects (both children and adults) with known or suspected primary immune disorders. We intend to characterize immune responsiveness to standard, well characterized antigens (vaccines) in subjects with primary immune disorders, and/or in subjects who have received treatments to correct their primary immune disorders. This will be an open label, prospective study investigating the functional status of the adaptive immune system. Up to 50 subjects may be enrolled. It is anticipated that subjects will be referred by any investigators at NIH studying inherited disorders of the immune system under their own protocols.

After giving standard vaccines, we will test specific antibody. The vaccines include licensed and universally mandated diphtheria and tetanus toxoid, two licensed pneumococcal vaccine formulations recommended for protection of children from pneumonia, and rabies vaccine licensed in 1997 (not the formerly available reaction-prone formulation). We will obtain peripheral blood samples from subjects before vaccination and at a specific time intervals after vaccination. Measurement of specific antibody titers will be conducted by the immunology laboratory at the Department of Laboratory Medicin at the NIH. Subjects may be offered one or more of the vaccines based on available information about their exposure history and their immune status, and the vaccines may be offered sequentially or in combination to shorten study time.

While the vaccines used here are often medically indicated and given outside of research protocols both to provide protection and to assess immune responses, the investigators have elected to use a protocol for the following reasons:

* Enhancement of subject understanding of the use of vaccines for in vivo assessment of immune responses.
* Emphasis on the importance of obtaining pre- and post-immunization blood samples to monitor how well the body's immune system is working.
* Administration of rabies vaccine to subjects who would not ordinarily need it.
* Recognition that vaccine side effects have been widely publicized and may be of concern to potential enrollees.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals being evaluated by NIH investigators for known or suspected primary immune disorders.

Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for at least 21 days prior to receipt of each vaccine and for the duration of study participation.

EXCLUSION CRITERIA:

Documented HIV infection.

Active malignancy.

Immunosuppressive therapy, other than steroids.

Symptomatic cardiac disease or ongoing treatment for it.

Pregnant or lactating women (due to restrictions on use of vaccines).

Surgery during the two weeks prior to entry.

Serious, ongoing, or uncontrolled infections.

Platelet count less than 40,000/microL or other coagulation disorder.

Any other major illness that, in the investigator's judgment, may substantially increase the risk associated with the patient's participation in this study.

History of previous systemic reaction to the particular vaccine product being considered for administration.

For RabAvert, persons known to be sensitive to:

* Processed bovine gelatin
* Chicken protein
* Neomycin
* Chlortetrycyline
* Amphotericin B

For Prevnar, persons with know or possible latex sensitivity.

The effects of the vaccines on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for at least 21 days prior to each vaccine and for the duration of study participation. Females of child bearing age will have a pregnancy test prior to each vaccination. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform study staff and her primary care physician immediately.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2002-06-13 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Post vaccine antibody level | 28 days
  To determine the function of T and B cells in vivo using immunizations in patients with known or suspected immune disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Gulbu Uzel, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-I-0226.html